CLINICAL TRIAL: NCT03588572
Title: A Randomized, Single Blind, Controlled, Longitudinal Study of the Effects of Venlafaxine Hydrochloride Capsules on the Language Function of Stroke Patients With Subcortical Aphasia Using fMRI
Brief Title: The Effect of Venlafaxine on Language Function in Patients With Subcortical Aphasia: A fMRI Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Yan Liu, Department director, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: LY-81471172
Record Dates: First submitted 2018-06-13; First posted 2018-07-17 (Actual); Results first posted 2019-10-03 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Subcortical Aphasia; Ischemic Stroke
Keywords: Behavioural evaluation; Functional magnetic resonance imaging; Venlafaxine
MeSH Terms: conditions — Ischemic Stroke | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Intervention Model Description: On the basis of conventional clinical treatment in both groups, the experimental group was given drug intervention, and the control group was not given drug treatment.
Who Masked: Participant
Masking Description: The investigator learned about the experimental grouping and medication situation, but the subjects did not know until the end of the experiment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venlafaxine Group (Experimental): The patients in venlafaxine group begin to take the venlafaxine hydrochloride capsules after the first visitation ( each containing venlafaxine 75mg), 1 capsule per day, until 4 weeks after randomization.
  Interventions: Drug: Venlafaxine hydrochloride capsules
- Controlled group (No Intervention): the patients in controlled group do not use the drug during the experiment, and the other treatments are same as the venlafaxine group.

INTERVENTIONS:
Drug: Venlafaxine hydrochloride capsules — The patients in venlafaxine group begin to take the venlafaxine hydrochloride capsules after the first visitation(the first day after randomization), each containing venlafaxine 75mg, 1 capsule per day, until 4 weeks after randomization
  Other Names: EFFEXOR XR®
  Arms: Venlafaxine Group

SUMMARY:
Previous studies have demonstrated that venlafaxine significantly improves the language function of healthy subjects and increase of fMRI activation in cortical language area. This study was designed to investigate the relationship between venlafaxine on the cortical language functional reorganization and clinical language improvements in the stroke patients with subcortical aphasia.

It is a randomized, controlled, single-blind, longitudinal trial which has approved by the ethics committee of Guangzhou General Hospital of Guangzhou Military Command, and all patients and their guardian should sign an informed consent. The patients will divide into the venlafaxine group and the control group according to the principle of randomization (random number table). The patients in the venlafaxine group begin to take a venlafaxine hydrochloride capsule after enrollment ( each containing venlafaxine 75mg), qd, until 4 weeks after randomization, and the control group do not. Assessments of language functional behavior and examines of functional magnetic resonance imaging (fMRI) should be performed on the first days (V1), 28±3 days (V2) and 90±3 days (V3) after randomization.

Through all this procession, we expect improve the language function of participants in experiment and clarify its mechanism,the research may help develop a new treatment for other patients with similar conditions.

DETAILED DESCRIPTION:
The cases will recruit from inpatients with acute ischemic stroke in Department of Cerebrovascular disease, The Guangzhou General Hospital of Guangzhou Military Command from June 2018 to June 2019. The diagnose of ischemic stroke is made using the diagnostic criteria of the International Association of Neurological Diseases and Stroke Association in 1982. The classification criteria for subcortical ischemic stroke are based on the current international TOAST etiological classification method.

It is a randomized, controlled, single-blind, longitudinal trial which has approved by the ethics committee of Guangzhou General Hospital of Guangzhou Military Command, and all patients and their guardian should sign an informed consent. The patients will divide into the venlafaxine group and the control group according to the principle of randomization (random number table). The patients in the venlafaxine group begin to take a venlafaxine hydrochloride capsule after enrollment ( each containing venlafaxine 75mg), qd, until 4 weeks after randomization, and the control group do not. Assessments of language functional behavior and examines of functional magnetic resonance imaging (fMRI) should be performed on the first days (Visit1,V1), 28±3 days (Visit2, V2) and 90±3 days (Visit3, V3) after randomization. Language functional behavioral assessments included the Chinese version of Western Aphasia Battery(WAB), spontaneous language frequency test(SLFT) and picture naming test(PNT). Examines of fMRI included task-state fMRI and resting-state fMRI. All patients received language rehabilitation training (twice a week, one hour each) which will be conducted by a professional rehabilitation physiotherapist from the Visitation1 until the end of Visitation3. The blood pressure and heart rate of each patient will be monitored and recorded on each visit, and two routine blood tests are performed at V0 and V3, including the blood routine and the liver and kidney function.

The test sample quantity is estimated using the sample size estimated by the professional software nQuery Advisor7.0. According to the main evaluation index of the effect of the previous literature on the efficacy of venlafaxine, the experimental group and the control group are 7.5±3.8 and 4.3±2.6，The standard deviation will be 3.26, and 0.05 will be the statistical meaning level (double tail). The test efficiency will be set to 0.83. The balance design will be used to estimate the sample size of the experimental group and the control group in 16 cases. In addition, considering the 20% missing rate, a total of 45 samples will be included in the study.

Task-state fMRI: an fMRI block design will be adopted, and DMDX software will be used to present each picture in series alternated between baseline (B) and activation (A) [B-A-B-A-B…]. Thirty-six animal pictures and 36 tool pictures accurately recognized by all subjects will be selected from the Snodgrass picture database. Six blocks of animal naming and six blocks of tool naming will be repeated, and each block continued for 18s with six pictures.the block-design diagram of picture naming task. The abstract figure of an American skunk which is unrecognized by all the subjects will be selected for baseline of animal naming. A schematic drawn arrow will be chosen for baseline picture of tool naming.Patients will be required to silently name the object in each picture without moving their lips. To avoid practice effects, the pictures used for activation will be different from those used in the behavioral evaluation. In the baseline phase, the participants will be asked to identify the orientation of the pictures by silently saying "upright" or "inverted." The subjects will receive task familiarization training prior to the test to ensure that there will be no substantive picture naming but only positional judgment in the baseline task.

Rest-state fMRI: During the rest-state fMRI scan, no task instruction will be given to the patient, and the patient will be completely relaxing, closing his eyes, breathing calmly, keeping his head still, but can not fall asleep, try to avoid any systematic thinking activities, scanning 8min.

Functional magnetic resonance data acquisition

The cranial brain scan will be performed using the US GE Signa HDx 3.0T Tesla superconducting magnetic resonance imaging system. The scanning sequence and parameters are as follows:

1. T1 structure imaging using FSPGR BRAVO sequence. The parameters included: time of repetition, 8.86 ms; time of echo, 3.52 ms; field of view, 24×24 cm2; in-plane resolution,256×256; slice thickness, 1 mm;interslice gap, 1 mm; and number of slices, 176.
2. Echo-Planar Imaging (EPI) is used to acquire task-state fMRI data.The parameters included: time of repetition, 3000ms; time of echo, 40 ms; field of view, 24×24 cm2; in-plane resolution,64×64; slice thickness, 4 mm; interslice gap, 1 mm; and number of slices, 34. Scan a sequence of 240s, a total of 12 min.
3. Echo-Planar Imaging (EPI) is used to acquire rest-state fMRI data.The parameters included: time of repetition, 3000ms; time of echo, 40 ms; field of view, 24×24 cm2; in-plane resolution,64×64; slice thickness, 4 mm; interslice gap, 1 mm; and number of slices, 34. A total of 8 min.

ELIGIBILITY:
Inclusion Criteria：

* The first stroke of the left single subcortical areas, within 72hours.
* Primary school or higher level,aged between 18-75, native language Chinese
* According to the commonly used eye chart examination, the corrected visual acuity is more than 1.0.
* According to the Edinburgh Handedness Questionnaire (EHQ) as the right handed.
* The language function was normal before the onset. After the onset, the language function was mildly to moderately impaired with Western Aphasia Battery (WAB) ( Aphasia Quotient (AQ) between in 60 to 88)
* The patient cooperate with the examination, they and their guardian signed the informed consent

Exclusion Criteria：

* History of organic diseases of the nervous system and history of craniocerebral trauma.
* History of epilepsy and psychosis.
* History of material dependence.
* Decompensation of important organ function.
* Hamilton Depression Scale(HAMD )>8 points.
* Hamilton Anxiety Scale(HAMA )>7 points.
* The Mini-Mental State Examination (MMSE)score <20 points.
* Dysphagia(difficult to take capsules).
* A history of allergens in component of venlafaxine.
* Pregnant women and breast-feeding women.
* Contraindication of MRI.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liu Yan, PhD, Study Chair — Guangzhou General Hospital of Guangzhou Military Command
Locations (2):
- China (2):
  - Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong
  - Cerebrovascular Department of General Hospital of Guangzhou Military Command of PLA, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pedersen PM, Jorgensen HS, Nakayama H, Raaschou HO, Olsen TS. Aphasia in acute stroke: incidence, determinants, and recovery. Ann Neurol. 1995 Oct;38(4):659-66. doi: 10.1002/ana.410380416. PMID 7574464
- [Background] Dickey L, Kagan A, Lindsay MP, Fang J, Rowland A, Black S. Incidence and profile of inpatient stroke-induced aphasia in Ontario, Canada. Arch Phys Med Rehabil. 2010 Feb;91(2):196-202. doi: 10.1016/j.apmr.2009.09.020. PMID 20159121
- [Background] Berthier ML. Poststroke aphasia : epidemiology, pathophysiology and treatment. Drugs Aging. 2005;22(2):163-82. doi: 10.2165/00002512-200522020-00006. PMID 15733022
- [Background] Engelter ST, Gostynski M, Papa S, Frei M, Born C, Ajdacic-Gross V, Gutzwiller F, Lyrer PA. Epidemiology of aphasia attributable to first ischemic stroke: incidence, severity, fluency, etiology, and thrombolysis. Stroke. 2006 Jun;37(6):1379-84. doi: 10.1161/01.STR.0000221815.64093.8c. Epub 2006 May 11. PMID 16690899
- [Background] Luria AR, Simernitskaya EG, Tubylevich B. The structure of psychological processes in relation to cerebral organization. Neuropsychologia. 1970 Jan;8(1):13-9. doi: 10.1016/0028-3932(70)90022-9. No abstract available. PMID 5522545
- [Background] Kim YH, You SH, Ko MH, Park JW, Lee KH, Jang SH, Yoo WK, Hallett M. Repetitive transcranial magnetic stimulation-induced corticomotor excitability and associated motor skill acquisition in chronic stroke. Stroke. 2006 Jun;37(6):1471-6. doi: 10.1161/01.STR.0000221233.55497.51. Epub 2006 May 4. PMID 16675743
- [Background] Debonnel G, Saint-Andre E, Hebert C, de Montigny C, Lavoie N, Blier P. Differential physiological effects of a low dose and high doses of venlafaxine in major depression. Int J Neuropsychopharmacol. 2007 Feb;10(1):51-61. doi: 10.1017/S1461145705006413. Epub 2006 May 11. PMID 16690006
- [Background] Berrocoso E, Mico JA. Role of serotonin 5-HT1A receptors in the antidepressant-like effect and the antinociceptive effect of venlafaxine in mice. Int J Neuropsychopharmacol. 2009 Feb;12(1):61-71. doi: 10.1017/S1461145708008766. Epub 2008 Apr 14. PMID 18405417
- [Background] Beique J, de Montigny C, Blier P, Debonnel G. Effects of sustained administration of the serotonin and norepinephrine reuptake inhibitor venlafaxine: II. In vitro studies in the rat. Neuropharmacology. 2000 Jul 24;39(10):1813-22. doi: 10.1016/s0028-3908(00)00018-6. PMID 10884562
- [Background] Thase ME, Entsuah AR, Rudolph RL. Remission rates during treatment with venlafaxine or selective serotonin reuptake inhibitors. Br J Psychiatry. 2001 Mar;178:234-41. doi: 10.1192/bjp.178.3.234. PMID 11230034
- [Background] Nemeroff CB, Entsuah R, Benattia I, Demitrack M, Sloan DM, Thase ME. Comprehensive analysis of remission (COMPARE) with venlafaxine versus SSRIs. Biol Psychiatry. 2008 Feb 15;63(4):424-34. doi: 10.1016/j.biopsych.2007.06.027. Epub 2007 Sep 24. PMID 17888885
- [Background] Thase ME, Entsuah R, Cantillon M, Kornstein SG. Relative antidepressant efficacy of venlafaxine and SSRIs: sex-age interactions. J Womens Health (Larchmt). 2005 Sep;14(7):609-16. doi: 10.1089/jwh.2005.14.609. PMID 16181017
- [Background] Schmitt AB, Bauer M, Volz HP, Moeller HJ, Jiang Q, Ninan PT, Loeschmann PA. Differential effects of venlafaxine in the treatment of major depressive disorder according to baseline severity. Eur Arch Psychiatry Clin Neurosci. 2009 Sep;259(6):329-39. doi: 10.1007/s00406-009-0003-7. Epub 2009 Mar 3. PMID 19255709
- [Background] Bauer M, Tharmanathan P, Volz HP, Moeller HJ, Freemantle N. The effect of venlafaxine compared with other antidepressants and placebo in the treatment of major depression: a meta-analysis. Eur Arch Psychiatry Clin Neurosci. 2009 Apr;259(3):172-85. doi: 10.1007/s00406-008-0849-0. Epub 2009 Jan 22. PMID 19165525
- [Background] Rickels K, Mangano R, Khan A. A double-blind, placebo-controlled study of a flexible dose of venlafaxine ER in adult outpatients with generalized social anxiety disorder. J Clin Psychopharmacol. 2004 Oct;24(5):488-96. doi: 10.1097/01.jcp.0000138764.31106.60. PMID 15349004
- [Background] Rudolph RL, Entsuah R, Chitra R. A meta-analysis of the effects of venlafaxine on anxiety associated with depression. J Clin Psychopharmacol. 1998 Apr;18(2):136-44. doi: 10.1097/00004714-199804000-00006. PMID 9555599
- [Background] Walker-Batson D, Curtis S, Natarajan R, Ford J, Dronkers N, Salmeron E, Lai J, Unwin DH. A double-blind, placebo-controlled study of the use of amphetamine in the treatment of aphasia. Stroke. 2001 Sep;32(9):2093-8. doi: 10.1161/hs0901.095720. PMID 11546902
- [Background] Feeney DM, Sutton RL. Pharmacotherapy for recovery of function after brain injury. Crit Rev Neurobiol. 1987;3(2):135-97. PMID 3107904
- [Background] Beversdorf DQ, Sharma UK, Phillips NN, Notestine MA, Slivka AP, Friedman NM, Schneider SL, Nagaraja HN, Hillier A. Effect of propranolol on naming in chronic Broca's aphasia with anomia. Neurocase. 2007 Aug;13(4):256-9. doi: 10.1080/13554790701595471. PMID 17886000
- [Background] Herrera-Guzman I, Herrera-Abarca JE, Gudayol-Ferre E, Herrera-Guzman D, Gomez-Carbajal L, Pena-Olvira M, Villuendas-Gonzalez E, Joan GO. Effects of selective serotonin reuptake and dual serotonergic-noradrenergic reuptake treatments on attention and executive functions in patients with major depressive disorder. Psychiatry Res. 2010 May 30;177(3):323-9. doi: 10.1016/j.psychres.2010.03.006. Epub 2010 Apr 10. PMID 20385412
- [Background] Fernandez B, Cardebat D, Demonet JF, Joseph PA, Mazaux JM, Barat M, Allard M. Functional MRI follow-up study of language processes in healthy subjects and during recovery in a case of aphasia. Stroke. 2004 Sep;35(9):2171-6. doi: 10.1161/01.STR.0000139323.76769.b0. Epub 2004 Aug 5. PMID 15297629
- [Background] Schweizer E, Thielen RJ, Frazer A. Venlafaxine:a novel antidepressant compound. Expert Opin Investig Drugs. 1997 Jan;6(1):65-78. doi: 10.1517/13543784.6.1.65. PMID 15989562
- [Background] Li CY, Song XZ, Han LX, Xie Q, Wang J, Li YK, Liu FD, Liu Y. The effects of venlafaxine on cortical motor area activity in healthy subjects: a pilot study. J Clin Psychopharmacol. 2014 Feb;34(1):93-8. doi: 10.1097/JCP.0000000000000056. PMID 24317453
- [Background] Xie Q, Liu Y, Li CY, Song XZ, Wang J, Han LX, Bai HM. The modulation of venlafaxine on cortical activation of language area in healthy subjects with fMRI study. Psychopharmacology (Berl). 2012 Oct;223(4):417-25. doi: 10.1007/s00213-012-2730-0. Epub 2012 May 4. PMID 22555622
- [Background] Adams HP Jr, Bendixen BH, Kappelle LJ, Biller J, Love BB, Gordon DL, Marsh EE 3rd. Classification of subtype of acute ischemic stroke. Definitions for use in a multicenter clinical trial. TOAST. Trial of Org 10172 in Acute Stroke Treatment. Stroke. 1993 Jan;24(1):35-41. doi: 10.1161/01.str.24.1.35. PMID 7678184
- [Background] Kertesz A. Western Aphasia Battery test manual. New York:NY: Grune & Stratton,1982.
- [Background] Hamilton M. Development of a rating scale for primary depressive illness. Br J Soc Clin Psychol. 1967 Dec;6(4):278-96. doi: 10.1111/j.2044-8260.1967.tb00530.x. No abstract available. PMID 6080235
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Damasio H, Grabowski TJ, Tranel D, Hichwa RD, Damasio AR. A neural basis for lexical retrieval. Nature. 1996 Apr 11;380(6574):499-505. doi: 10.1038/380499a0. PMID 8606767
- [Background] Kim H, Na DL. Normative data on the Korean version of the Western Aphasia Battery. J Clin Exp Neuropsychol. 2004 Nov;26(8):1011-20. doi: 10.1080/13803390490515397. PMID 15590457
- [Background] Berthier ML, Pulvermuller F, Davila G, Casares NG, Gutierrez A. Drug therapy of post-stroke aphasia: a review of current evidence. Neuropsychol Rev. 2011 Sep;21(3):302-17. doi: 10.1007/s11065-011-9177-7. Epub 2011 Aug 16. PMID 21845354

RESULTS

PARTICIPANT FLOW:
Period: Visitation 1
Arm/Group | Venlafaxine Group | Controlled Group
Started | 22 | 21
Completed | 21 | 20
Not Completed | 1 | 1
Not completed — Lack of Efficacy | 1 | 1
Period: Visitation 2
Arm/Group | Venlafaxine Group | Controlled Group
Started | 21 | 20
Completed | 19 | 18
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Visitation 3
Arm/Group | Venlafaxine Group | Controlled Group
Started | 19 | 18
Completed | 16 | 16
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Venlafaxine Group | Controlled Group | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 55.19 (10.94) | 54.06 (9.00) | 54.62 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 9 | 11 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 16 | 16 | 32
Body Mass Index（BMI） [Mean (Standard Deviation); unit: kg/m^2] | 23.28 (1.20) | 23.15 (1.31) | 23.22 (1.24)
Education Level [Mean (Standard Deviation); unit: years] | 8.63 (3.07) | 8.44 (2.25) | 8.54 (2.77)
Vascular Risk Factors（Hypertension, Diabetes, Hyperlipidemia, Smoking） [Count of Participants; unit: Participants]
  Hypertension: Yes | 12 | 13 | 25
  Hypertension: No | 4 | 3 | 7
  Diabetes: Yes | 3 | 4 | 7
  Diabetes: No | 13 | 12 | 25
  Hyperlipidemia: Yes | 7 | 8 | 15
  Hyperlipidemia: No | 9 | 8 | 17
  Smoking: Yes | 6 | 7 | 13
  Smoking: No | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: A Change of Outcome Measure:the Chinese Version of Western Aphasia Battery(WAB)
Description: The main outcome measure for this scale is Aphasia Quotient(AQ) which mainly tests the ability of spontaneous speech, oral comprehension, repetition, and naming, and reflects the severity of aphasia, and can be used as a reliable indicator to evaluate the improvement and deterioration of aphasia. Score fluctuation is 0-100 points, the normal value is 98.4-100 points, AQ<93.8 can be judged as language dysfunction.
Time Frame: This is an outcome measure to assess the improvement of language function from onset to 3 months after treatment. Thus, participates will undergo this assessment on the first days (V1), 28±3 days (V2), and 90±3 days (V3) after randomization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venlafaxine Group | Controlled Group
Number analyzed (Participants) | 16 | 16
score on a scale
  Visitation 1 | 78.16 (7.93) | 78.60 (6.38)
  Visitation 2 | 88.24 (6.15) | 83.51 (5.37)
  Visitation 3 | 94.23 (4.38) | 88.55 (3.95)

2. Secondary Outcome: A Change of Outcome Measure:Spontaneous Language Frequency Test(SLFT)
Description: This test mainly assesses spontaneous speech fluency of participants.It requires participants name as many food names as possible within one minute, and each correct one to give one point.The higher the score, the better the language function.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venlafaxine Group | Controlled Group
Number analyzed (Participants) | 16 | 16
score on a scale
  Visitation 1 | 5.31 (1.99) | 5.75 (1.81)
  Visitation 2 | 9.31 (1.54) | 8.13 (1.5)
  Visitation 3 | 12.69 (1.49) | 10.81 (1.33)

3. Secondary Outcome: A Change of Outcome Measure:Picture Naming Test(PNT)
Description: This test mainly assesses the ability of picture name of participants.we used a program for displaying named pictures on a computer screen (60 photos in total, of which 20 were Chinese celebrity faces). Each image was displayed in 3 seconds, and 1 point was correctly named for an image.The faces of celebrities were selected from the picture database of Chinese celebrities in the State Key Laboratory of Cognitive Neuroscience and Learning at Beijing Normal University.Score fluctuation is 0-60 points, the higher the score, the better the ability of picture name.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venlafaxine Group | Controlled Group
Number analyzed (Participants) | 16 | 16
score on a scale
  Visitation 1 | 39.19 (5.19) | 38.31 (5.23)
  Visitation 2 | 46.75 (4.36) | 43.31 (4.45)
  Visitation 3 | 52.25 (2.6) | 48.31 (3.96)

4. Secondary Outcome: Follow-up Measurement: Hamilton Depression Rating Scale (HAMD)
Description: The Hamilton Depression Rating Scale (HAMD) has proven useful for many years as a way of determining a patient's level of depression before, during, and after treatment. It generally takes 15-20 minutes to complete the interview and score the results. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine items are scored from 0-2. HAMD Scoring Instructions:0-7=Normal, 8-13 = Mild Depression, 14-18 = Moderate Depression, 19-22 = Severe Depression, ≥ 23 = Very Severe Depression(i.e.,Minimum 0 points and maximum 50 points, the higher the score, the greater the likelihood of depression).
Time Frame: We must determine that the participant is not in depression at each follow-up. Thus, participates will undergo this assessment on the first days (V1), 28±3 days (V2), and 90±3 days (V3) after randomization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venlafaxine Group | Controlled Group
Number analyzed (Participants) | 16 | 16
score on a scale
  Visitation 1 | 5.63 (0.96) | 5.25 (0.93)
  Visitation 2 | 4.94 (0.57) | 4.63 (0.81)
  Visitation 3 | 4.06 (0.93) | 3.88 (0.72)

5. Secondary Outcome: Follow-up Measurement: Hamilton Anxiety Rating Scale (HAMA)
Description: The Hamilton Anxiety Rating Scale (HAMA) is a widely used and well-validated tool for measuring the severity of a patient's anxiety. The HAMA is composed of 14 items and takes 15-20 minutes to complete the interview and score the results. Each item is scored on a 5-point scale, ranging from 0=not present to 4=severe.HAMA Scoring Instructions:0-8=Normal, 8-13= Possible Anxiety, 14-17 = Mild Anxiety, 18-24 = Moderate Anxiety, 25-30 = Severe Anxiety(i.e.,the higher the score, the greater the likelihood of anxiety).
Time Frame: We must determine that the participant is not in anxiety at each follow-up. Thus, participates will undergo this assessment on the first days (V1), 28±3 days (V2), and 90±3 days (V3) after randomization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venlafaxine Group | Controlled Group
Number analyzed (Participants) | 16 | 16
score on a scale
  Visitation 1 | 4.88 (0.89) | 4.63 (1.09)
  Visitation 2 | 4.13 (0.96) | 4.00 (0.73)
  Visitation 3 | 3.56 (0.89) | 3.25 (0.78)

6. Secondary Outcome: Follow-up Measurement: Mini-Mental State Examination (MMSE)
Description: The Mini-Mental State Examination (MMSE) is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. Administration of the test takes between 5 and 10 minutes. The MMSE test includes simple questions and problems in a number of areas: the time and place of the test, repeating lists of words, arithmetic such as the serial sevens, language use and comprehension, and basic motor skills. Any score greater than or equal to 24 points (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.The raw score may also need to be corrected for educational attainment and age.
Time Frame: We must determine that the participant is not in moderate or more cognitive impairment at each follow-up. Thus, participates will undergo this assessment on the first days (V1), 28±3 days (V2), and 90±3 days (V3) after randomization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venlafaxine Group | Controlled Group
Number analyzed (Participants) | 16 | 16
score on a scale
  Visitation 1 | 23.81 (1.22) | 23.88 (1.15)
  Visitation 2 | 25.38 (0.96) | 25.00 (1.03)
  Visitation 3 | 26.38 (0.81) | 26.19 (0.83)

ADVERSE EVENTS:
Time Frame: 1 year
Description: We will collect medical history and physical examination results of participates, We use various indicators to identify adverse events，e.g., blood routine, urine routine, stool routine, liver and kidney function examination.
Arm/Group | Venlafaxine Group | Controlled Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT03588572/Prot_002.pdf
  • Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT03588572/SAP_003.pdf